CLINICAL TRIAL: NCT06882200
Title: Benefit of the Bathysmed® Diving Protocol on Emotional Eating in Obese Patients: A Prospective Randomized Study
Brief Title: A Combined Mindfulness-diving Protocol on Emotional Eating in Obese Patients: A Prospective Randomized Study
Acronym: OBEDIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BATHYSMED (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BTY-2022-05-OBEDIVE; 4021591/1 (Other Grant/Funding Number: BPI France)
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Obesity and Overweight
Keywords: obesity; mindfulness; diving; exercise
MeSH Terms: conditions — Obesity; Overweight; Motor Activity | interventions — Primary Health Care; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diving group (Experimental): The program included ten scuba-diving sessions with mindfulness training, twice a week for five weeks, alongside standard care for obesity in a primary care centre in Montpellier
  Interventions: Other: A combined mindfulness and therapeutic scuba-diving protocol
- Control group (Placebo Comparator): Standard care included regular appointments and health education with their general practitioner and monthly appointments with the dietician and psychotherapist at the primary care centre in Montpellier, France throughout the study.
  Interventions: Other: Control group regular follow up in primary care

INTERVENTIONS:
Other: A combined mindfulness and therapeutic scuba-diving protocol — The Bathysmed program is a unique scuba diving program that combines scuba immersion with techniques from mindfulness meditation, psychology and sports mental preparation. The program includes 30 different exercises over ten scuba-diving sessions with mindfulness training, twice a week for five weeks.
  Other Names: BathysMed Diving protocol
  Arms: Diving group
Other: Control group regular follow up in primary care — Standard care includes regular appointments and health education with their general practitioner and monthly appointments with the dietician and psychotherapist at the primary care centre in Montpellier, France throughout the study. This care includes monthly sessions on diet, exercise and general stress management with a registered dietician.
  Other Names: Control group
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to learn if a combined minfulness-diving program has an impact on emotional eating in adults with obesity. The main questions it aims to answer are:

Does the BathysMed protocol have an impact on emotional eating after the 2 months diving protocol? Researchers will compare the diving program to a control group of adult patients with obesity.

Participants will be asked to participate in the combined mindfulness-diving protocol for 2 months, and complete the questionnaires at baseline, 2, 5, and 8 months follow up.

DETAILED DESCRIPTION:
This unblinded randomized controlled trial is performed in the community setting, Montpellier, France. Adults with a BMI > 30kg/m2 were randomly assigned (1:1) to a Bathysmed® 2-month program (intervention group) therapeutic scuba-diving protocol with mindfulness exercises plus standard care, or stand-alone standard care including dietary and psychological support (control group). The primary outcome was the mean change in the emotional eating subscale of the Dutch Eating Behaviour Questionnaire (DEBQ-EE) at 2-months as intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* patients with obesity (Body Mass Index BMI > 30kg/m2),
* adults over the age of 18 able to provide written consent
* affiliated to public medical insurance.

Exclusion Criteria:

* BMI > 45 kg/m2,
* older than 60 years,
* unable to walk,
* known psychiatric pathology apart from anxiety and depression,
* intellectual deficit,
* routinely practising meditation,
* a known contra-indication to scuba-diving
* known past medical history of cardiac problems.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
DEBQ-EE | 2 months
  The primary outcome was the mean change in the emotional eating subscale of the Dutch Eating Behaviour Questionnaire (DEBQ-EE) at the end of the two-month protocol.

SECONDARY OUTCOMES:
DEBQ-EE at 5 and 8 months follow up | 5 and 8 months follow up
  emotional eating subscale of the Dutch Eating Behaviour Questionnaire (DEBQ-EE) at 5 and 8 months follow up
DEBQ-RE | 2, 5 and 8 months follow up
  Change in the Restrictive eating subscale of the Dutch Eating Behaviour Questionnaire (DEBQ-EE) between baseline and two, five and eight months follow up
DEBQ-ExtE | 2, 5 and 8 months follow up
  Change in the external eating subscale of the Dutch Eating Behaviour Questionnaire (DEBQ-EE) between baseline two, five and eight months follow up
WSSQ | 2, 5 and 8 months follow up
  Change in weight bias internalisation (WBI) and weight self-stigma using the Weight Self Stigma Questionnaire (WSSQ), score between baseline and 2, 5 and 8 months follow up
EQVOD scale | 2, 5 and 8 months follow up
  Change in the quality of life using a specific questionnaire for obese patients EQVOD (l'échelle de Qualité de Vie Obésité et Diététique) (17); between baseline and 2 , 5 and 8 months follow up
PSS Score | 2, 5 and 8 months follow up
  Evaluation of Perceived Stress Scale of Cohen score (PSS), between baseline and 2, 5 and 8 months follow up
Weight (kg) | 2, 5 and 8 months follow up
  Weight measured in Kg
BMI kg/m2 | 2, 5 and 8 months follow up
  BMI kg/m2 Body Mass Index
Waist circumference | 2, 5 and 8 months follow up
  Waist circumference (cm)

CONTACTS AND LOCATIONS:
Locations (1):
- BathysMed, Montpellier, France

IPD SHARING:
Plan to Share IPD: Yes